CLINICAL TRIAL: NCT04051645
Title: Problems of Measurement and Evaluation of Breathing Effort in Spontaneously Breathing Subjects
Brief Title: Evaluation of Breathing Effort in Spontaneously Breathing Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: iWoBvsiPTP
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Work of breathing; Pressure Time Product; imposed WoB; imposed PTP; flow resistance

STUDY DESIGN:
Intervention Model Description: In the experiment, the proband will breathe through the D-Lite measuring screen of the Datex-Ohmeda S/5 Patient Monitor patient monitor (GE, USA). Unlike clinical practice, an adjustable flow resistance will be connected to the system. The flow resistance is set by adjustable by a removable diaphragm with different hole diameters according to the intended flow resistance.
Masking Description: No masking will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing through a system with adjustable flow resistance (Experimental): During the experiment, the volunteers will breathe through ten adjustable flow resistances and their work of breathing will be measured.
  Interventions: Device: Breathing through a system with adjustable flow resistance

INTERVENTIONS:
Device: Breathing through a system with adjustable flow resistance — The proband will breathe through the adjustable flow resistance within the experiment, to which a standard D-lite Flow sensor will be connected, and the airway pressure, flow, minute consumption, oxygen and carbon dioxide, tidal volume, oxygen saturation of peripheral blood and oxygen and carbon dioxide concentrations in both inspired and expired air will be recorded using the Datex-Ohmeda S/5 Patient Monitor vital signs monitor.
  The proband will breathe through the flow resistors in a randomized order, and pre-defined three-minute pauses will be maintained between measurements with different flow resistance values. Each measurement will take approximately two minutes and will be measured on ten different flow resistances.

SUMMARY:
The aim of the research project is to evaluate the breathing effort using the Work of Breathing (WoB) and Pressure-Time Product (PTP) parameters, depending on the increasing flow resistance. The research project is concerned with assessing the increased (imposed) breathing effort using the Work of Breathing (iWoB) and the Pressure-Time Product (iPTP).

The main hypothesis tested is the differential effect of flow resistance on iWoB and iPTP parameters in spontaneous breathing of healthy probands.

DETAILED DESCRIPTION:
Due to the different calculation of iWoB and iWoB, these parameters may be affected at higher flow resistance values. The proposed experiment will be used to compare iWoB and iPTP obtained during spontaneous breathing to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females > 18 and < 40 years old
* Signed informed consent has been obtained

Exclusion Criteria:

* Respiratory disease
* Pregnancy
* Cardiovascular disease
* Diabetes mellitus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
iWoB | through study completion, an average of 1 year
  imposed work of breathing in J/s/L
iPTP | through study completion, an average of 1 year
  imposed pressure time product in Pa.s/L

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Prof., Study Director — Czech Technical University in Prague, Fac. of Biomedical Engineering
Locations (1):
- Department of Biomedical Technology Faculty of Biomedical Engineering Czech Technical University in Prague, Kladno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
Anonymous data from anesthesia monitor of vital functions

REFERENCES:
- [Background] Bellani G, Pesenti A. Assessing effort and work of breathing. Curr Opin Crit Care. 2014 Jun;20(3):352-8. doi: 10.1097/MCC.0000000000000089. PMID 24722059
- [Background] de Vries H, Jonkman A, Shi ZH, Spoelstra-de Man A, Heunks L. Assessing breathing effort in mechanical ventilation: physiology and clinical implications. Ann Transl Med. 2018 Oct;6(19):387. doi: 10.21037/atm.2018.05.53. PMID 30460261
- [Background] Dodd DS, Kelly S, Collett PW, Engel LA. Pressure-time product, work rate, and endurance during resistive breathing in humans. J Appl Physiol (1985). 1988 Apr;64(4):1397-404. doi: 10.1152/jappl.1988.64.4.1397. PMID 3378975
- [Background] Collett PW, Perry C, Engel LA. Pressure-time product, flow, and oxygen cost of resistive breathing in humans. J Appl Physiol (1985). 1985 Apr;58(4):1263-72. doi: 10.1152/jappl.1985.58.4.1263. PMID 3988680
- [Background] Cabello B, Mancebo J. Work of breathing. Intensive Care Med. 2006 Sep;32(9):1311-4. doi: 10.1007/s00134-006-0278-3. Epub 2006 Jul 13. No abstract available. PMID 16838150